CLINICAL TRIAL: NCT06320080
Title: Phase Ib Clinical Study Evaluating the Efficacy and Safety of TQB2223 Injection Combined With Penpulimab Injection in the Treatment of Advanced Hepatocellular Carcinoma
Brief Title: Clinical Study of TQB2223 Injection Combined With AK105 Injection in the Treatment of Advanced Hepatocellular Carcinoma.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was closed due to business reasons. Closure was not prompted by any safety or efficacy concerns.
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2223-AK105-Ib-01
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2024-11

CONDITIONS: Advanced Hepatocellular Carcinoma
MeSH Terms: interventions — penpulimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2223 injection+ AK105 Injection (Experimental): TQB2223 injection combined with AK105 (Penpulimab) injection, once every three weeks. 21 days as a treatment cycle.
  Interventions: Drug: TQB2223 injection; Drug: Penpulimab Injection

INTERVENTIONS:
Drug: TQB2223 injection — TQB2223 is an anti- lymphocyte activation gene-3 (LAG-3) antibody.
Drug: Penpulimab Injection — Penpulimab Injection is an anti programmed death-1 (PD-1) antibody.

SUMMARY:
TQB2223 is a recombinant, fully human antibody that binds to lymphocyte activation gene-3 (LAG-3) and blocks the LAG-3/ major histocompatibility complex class II (MHC-II) interaction, thus allowing for increased T-cell proliferation and cytokine production. This is a phase Ib study aimed at evaluating the safety, tolerability, and immunogenicity characteristics of TQB2223 injection combined with AK105 injection in the treatment of advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years old, an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1, and life expectancy ≥3 months;
* Hepatocellular carcinoma (HCC) patients confirmed by pathological histology or cytology examination or meeting the clinical diagnostic criteria for hepatocellular carcinoma according to the American Association for the Study of Liver Diseases (AASLD) or the Diagnosis and Treatment Guidelines for Primary Liver Cancer (2022 edition);
* Have not received any immunotherapy for advanced HCC previously;
* Subjects with a China liver cancer staging (CNLC) of stage III [or Barcelona clinical staging of liver cancer (BCLC) of stage C], or CNLC-II (BCLC-B) subjects who are not suitable for local treatment (such as hepatic artery chemotherapy and embolization) and surgical treatment, or cannot benefit from local treatment and surgical treatment as determined by the investigators;
* Child Pugh liver function grading: Grade A or B (≤ 7 points)
* Subjects with advanced malignant tumors who failed standard treatment or lacked effective treatment;
* The main organs function well;
* Male or female patient had no plans to become pregnant and agree to voluntarily take effective contraceptive measures during the study to at least 6 months after the last dose of study drug.

Exclusion Criteria:

* Concurrent secondary malignancy or other malignancy with no evidence of disease within 5 years prior to the first dose;
* Within 28 days prior to the first dose, received significant surgical treatment, or with obvious traumatic injury or long-term unhealed wound or fracture;
* Patients who experienced any bleeding or bleeding events ≥ CTC AE level 3 within 4 weeks prior to the first dose; Individuals who have experienced arterial/venous thrombosis events within 6 months prior to the first dose, such as cerebrovascular accidents, deep vein thrombosis, and pulmonary embolism; Low molecular weight heparin treatment is allowed, and antiplatelet drugs are prohibited throughout the entire study period;
* A history of gastrointestinal bleeding such as active gastric and duodenal ulcers, persistent positive fecal occult blood, and ulcerative colitis within 6 months prior to the first dose; Or other conditions determined by investigators that may cause gastrointestinal bleeding or perforation;
* Patients with portal hypertension and at high risk of bleeding considered by the investigators, or have been confirmed by gastroscopy to have red signs or severe esophageal and gastric varicose veins.
* Individuals with a history of psychiatric drug abuse who are unable to quit or have mental disorders;
* Individuals who have previously received or are preparing to undergo allogeneic bone marrow transplantation or solid organ transplantation within 6 months;
* History of hepatic encephalopathy;
* History of uncontrolled intercurrent illness;
* Participants who have participated in other clinical trials of anti-tumor drugs and used other investigational anti-tumor drugs within 4 weeks prior to the first dose;
* Unstable or serious concurrent medical conditions, as assessed by the Investigators, that would substantially increase the risk-benefit ratio of participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From date of the first dose until the date of first documented progression or date of death from any cause, assessed up to 100 weeks.
  The percentage of subjects with Complete Response (CR) or partial response (PR) assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 and Immune-Modified Response Evaluation Criteria In Solid Tumors (iRECIST).
Progression-free survival (PFS) | From date of the first dose until the date of first documented progression or date of death from any cause, assessed up to 100 weeks
  The time from the first dose of TQB2223 to the first occurrence of disease progression or death from any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | From date of the first dose until the date of first documented progression or date of death from any cause, assessed up to 100 weeks
  The time from the first treatment to death from any cause.
Disease control rate (DCR) | From date of the first dose until the date of first documented progression or date of death from any cause, assessed up to 100 weeks
  The proportion of subjects with Complete response (CR), Partial response (PR), or Stable Disease (SD).
Duration of Response (DOR) | From date of the first dose until the date of first documented progression or date of death from any cause, assessed up to 100 weeks
  The time from first documented response to documented disease progression or death.
Number of patients with adverse events (AEs) and/or serious adverse events (SAEs) | From the time of informed consent to 28 days after the last dose
  Assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Immunogenicity | within 1 hour before dose in the 1st, 2nd, 4th, and 8th cycle. 30 and 90 days after the last dose. 21 days as a treatment cycle.
  The occurence of Anti-drug antibody (ADA) after administration

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Affiliated Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Hubei Provincial Tumor Hospital, Wuhan, Hubei
  - Hunan Provincial Tumor Hospital, Changsha, Hunan